CLINICAL TRIAL: NCT06749457
Title: A Phase I/IIa Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of AZD7760 in Healthy Participants and in Patients With End-stage Kidney Disease Receiving Hemodialysis Through a Central Venous Catheter
Brief Title: A Study to Evaluate AZD7760 Safety and Pharmacokinetics in Healthy Adults (Phase I) and Adults With End-stage Kidney Disease on Hemodialysis With a Central Venous Catheter (Phase IIa)
Acronym: PEAK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D7480C00001
Record Dates: First submitted 2024-12-23; First posted 2024-12-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Staphylococcus Aureus
Keywords: Bloodstream infection; End-stage kidney disease
MeSH Terms: conditions — Staphylococcal Infections; Sepsis; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase I: AZD7760 Dose A (Experimental): Participants will receive a single dose of AZD7760 Dose A intravenously on Day 1.
  Interventions: Drug: AZD7760
- Phase I: AZD7760 Dose B (Experimental): Participants will receive a single dose of AZD7760 Dose B intravenously on Day 1.
  Interventions: Drug: AZD7760
- Phase I: AZD7760 Dose C (Experimental): Participants will receive a single dose of AZD7760 Dose C intravenously on Day 1.
  Interventions: Drug: AZD7760
- Phase I: Placebo (Placebo Comparator): Participants will receive a single dose of placebo on Day 1.
  Interventions: Other: Placebo
- Phase IIa: AZD7760 Dose D and Placebo (Experimental): Participants will receive AZD7760 Dose D and placebo on Day 1 on Day 91.
  Interventions: Drug: AZD7760; Other: Placebo
- Phase IIa: AZD7760 Dose E (Experimental): Participants will receive AZD7760 Dose E on Day 1 and Day 91.
  Interventions: Drug: AZD7760
- Phase IIa: Placebo (Placebo Comparator): Participants will receive placebo on Day 1 and on Day 91.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD7760 — Participants will receive AZD7760 as a single intravenous infusion.
  Arms: Phase I: AZD7760 Dose A; Phase I: AZD7760 Dose B; Phase I: AZD7760 Dose C; Phase IIa: AZD7760 Dose D and Placebo; Phase IIa: AZD7760 Dose E
Other: Placebo — Participants will be administered placebo through intravenous infusion.
  Arms: Phase I: Placebo; Phase IIa: AZD7760 Dose D and Placebo; Phase IIa: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (PK) of AZD7760 when given as an intravenous infusion to healthy participants (Phase I) or participants with end-stage kidney disease receiving hemodialysis through a central venous catheter (Phase IIa).

DETAILED DESCRIPTION:
In the Phase I portion of the study, participants will be randomized to receive one of 3 dosages of AZD7760 or placebo as a single intravenous infusion.

Study details include:

* A 28-day Screening Period.
* A Dosing Period of 3 days in which a single intravenous infusion will be given on Day 1.
* A Follow-up Period of 12 months from the time of administration of the study intervention.

In the Phase IIa portion of the study, participants will be randomized to receive either AZD7760 or placebo as 2 intravenous infusions given 3 months apart.

Study details include:

* A 28-day Screening Period.
* A Dosing Period in which 2 intravenous infusions will be given 3 months apart (Day 1 and Day 91).
* A Follow-up Period of 12 months after the last administration of the study intervention on Day 91.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

* Participant must be 18 to 55 years of age (inclusive), at the time of signing the informed consent.
* Body weight ≥ 45 kilograms (kg) and ≤ 110 kg and Body Mass Index (BMI) within the range ≥ 18.0 to ≤ 30.0 kilograms per square meter (kg/m2) (inclusive) at screening.
* Healthy participants with no clinically significant concomitant diseases or medications (except for those specifically permitted by the protocol) according to medical history, physical examination, screening safety laboratory tests, and screening parameters, as perthe judgement of the investigator.

Phase IIa:

* Participant must be ≥ 18 years of age at the time of signing the informed consent.
* Participants who meet all of the following disease status requirements:

  1. Diagnosed with End-stage kidney disease (ESKD).
  2. Requiring hemodialysis through a tunneled central venous catheter as the primary vascular access for hemodialysis.
  3. Receiving hemodialysis for treatment of ESKD for at least 90 days before randomization.
  4. At least 3 previous dialysis sessions using current dialyzer.
  5. Receiving adequate hemodialysis based on a single-pool Kt/V measurement > 1.2 within the last 30 days.
  6. No new medications have been added to the participant's regimen in the last 2 weeks prior to dosing. 'New medication' is defined as any medication that has not been prescribed or used by the participant previously (including formulation changes). Medication previously prescribed or used by the participant with dose adjustments is allowed and not considered as new medication for the purpose of this study.
  7. Not taking long-term systemic antibiotics with activity against S aureus.

Exclusion Criteria:

Phase I:

* Known hypersensitivity to any component of the study intervention
* Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of monoclonal antibodies (mAbs).
* Clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
* Aspartate Aminotransferase (AST) or alanine Aminotransferase (ALT) above 1.5 × upper limit of normal (ULN) at screening. Testing may be repeated once at the investigator's discretion.
* Estimated glomerular filtration rate < 90 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration equation at screening.
* Hemoglobin or platelet count below the lower limit of normal at screening. Testing may be repeated once at the investigator's discretion.
* White blood cell counts outside normal reference ranges unless judged by the investigator to be out of range given the known variation in white blood cell count reference interval by ethnicity. Testing may be repeated once at the investigator's discretion.
* History of malignancy other than treated non-melanoma skin cancers or locally treated cervical cancer in the previous 5 years.
* Any laboratory value in the screening panel that, in the opinion of the investigator, is clinically significant or might confound analysis of study results. Testing may be repeated once at the investigator's discretion.
* Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening, as judged by the investigator.
* Acute (time-limited) illness, including fever ≥ 38 °C (100.4 °F), one day prior to or on day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves within the 28-day Screening Period or may be rescreened once.
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening.
* Any condition that has the potential to increase clearance of the study intervention (eg, protein loss conditions such as severe enteropathies, or plasmapheresis).
* Blood drawn in excess of a total of 450 milliliters (mL) (1 unit) for any reason within 2 months prior to screening.
* Absence of suitable veins for blood sampling and administration of study intervention.
* Any other condition that would compromise safety of the participants.
* Any condition that, in the opinion of the investigator, might interfere with evaluation of the study intervention or interpretation of participant safety or study results.

Phase IIa:

* Known hypersensitivity to any component of the study intervention.
* History of allergic disease or reactions likely to be exacerbated by any component of the study intervention as listed in dose formulation section.
* Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of mAbs.
* Hemoglobin < 9 g/dL at screening considered by the investigator to be due to acute condition(s). Testing may be repeated once at the investigator's discretion.
* Serum albumin of < 3 g/dL at screening considered by the investigator to be due to acute condition(s). Testing may be repeated once at the investigator's discretion.
* Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thrombotic/thromboembolic event (eg, deep vein thrombosis or pulmonary embolism, but excluding vascular access thrombosis) within 90 days prior to randomization.
* Known S aureus infection within 90 days of study entry.
* Known acute viral or bacterial infection or symptoms/signs consistent with such an infection within the 21 days prior to infusion or study intervention. Mild intercurrent viral illness with a temperature of 38.1 °C (100.6 °F) or less does not require exclusion, if in the judgement of the investigator this illness will not interfere with the evaluation of the mAb.
* Participants with malignancy undergoing chemotherapy.
* Scheduled date for living donor kidney transplant.
* Plans to switch to peritoneal dialysis within the primary endpoint time period (181 days).
* Participants with a scheduled calendar date for transition to arteriovenous graft or arteriovenous graft in place and maturing.
* Participants with a scheduled calendar date for transition to arteriovenous fistula, or arteriovenous fistula in place and maturing, with anticipated use of fistula within 90 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 231 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: Occurence of adverse events (AEs) | Day 1 to Day 181
  To evaluate the safety of AZD7760 administered as a single intravenous (IV) Dose A, B, or C.
Phase I: Occurence of medically-attended adverse events (MAAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) | Day 1 to Day 361
  To evaluate the safety of AZD7760 administered as a single IV Dose A, B, or C.
Phase IIa: Occurrence of AEs, MAAEs, SAEs, and AESIs | Day 1 to Day 181
  To evaluate the safety of AZD7760 compared with placebo as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E

SECONDARY OUTCOMES:
Phase I: Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 to Day 361
  To characterize the pharmacokinetics (PK) of AZD7760 in serum.
Phase I: Time to reach peak or maximum observed concentration following drug administration (tmax) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Area under plasma concentration-time curve from zero extrapolated to infinity (AUCinf) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Apparent volume of distribution at steady state (Vss) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Apparent volume of distribution at the terminal phase (Vz) | Day 1 to Day 361
  To characterize the PK of AZD7760 in serum.
Phase I: Incidence of ADA | Day 1 to Day 361
  To evaluate ADA responses to AZD7760 in serum.
Phase IIa: Cmax | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: tmax | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: t1/2λz | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: AUClast | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: AUCinf | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: Vss | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: Vz | Day 181 to Day 451
  To characterize the serum PK profiles of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: Incidence of anti-drug antibodies (ADAs) to AZD7760 in serum | Day 181 to Day 451
  To evaluate ADA responses to AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: Occurrence of AEs | Day 1 to Day 181
  To evaluate the safety to Day 181 of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E
Phase IIa: Occurrence of MAAEs, SAEs, and AESIs | Day 1 to Day 451
  To evaluate the safety to Day 451 of AZD7760 administered as:
  * A single IV dose (at Day 1) of Dose D followed by placebo (at Day 91)
  * 2 IV doses (at Day 1 and Day 91) of Dose E

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Research Site, Huntsville, Alabama
  - Research Site, Chula Vista, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oxnard, California
  - Research Site, Riverside, California
  - Research Site, San Dimas, California
  - Research Site, Tarzana, California
  - Research Site, Valencia, California
  - Research Site, Victorville, California
  - Research Site, Englewood, Colorado
  - Research Site, Bradenton, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Jersey City, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Ridgewood, New York
  - Research Site, Kinston, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/